CLINICAL TRIAL: NCT02526433
Title: The Impact of Creative Interventions on Symptoms of Postnatal Depression (Cohort Study)
Status: Completed | Type: Observational
Sponsor: Royal College of Music (Other)
Collaborators: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: SATB2015b
Record Dates: First submitted 2015-08-14; First posted 2015-08-18 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Depression, Postpartum
Keywords: depression; mental wellbeing; motherhood; music; alternative therapies
MeSH Terms: conditions — Depression, Postpartum; Depression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pregnancy women and new mothers: The study tracks what interventions women are already registered in and compares these with their mental wellbeing.

SUMMARY:
Post-natal depression (PND) is anticipated to affect 12.9% of new mothers with at least 75,000 cases per year in the UK alone. However, despite this, there is currently a worrying lack of support for new mothers, with data suggesting that 64% of healthcare trusts in the UK do not have a strategy for treating PND, and flaws in the current pharmacological and psychological treatment models. Consequently, research into promising psychosocial interventions such as music is critical to developing new paradigms for treating PND.

This project is an ambitious programme of research that investigates links between the mental health of women in the later stages of pregnancy and first 9 months post birth and their use of psychosocial interventions including music.

DETAILED DESCRIPTION:
The study uses an online questionnaire to achieve a cross-sectional view of the mental health of women across England in the final stages of pregnancy and the first 9 months post birth, how much and in what ways music is used by these women, and whether there are any associations between music and mental health. The study aims to recruit between 1,000 and 5,000 women to take the anonymous questionnaire. However, women who complete the questionnaire while still pregnant will be invited to complete three further questionnaires shortly post-birth and 3 months later to gather longitudinal data to analyse change across pregnancy into post-birth (aiming for 500 of the 1,000 undertaking this repeated measurement).

Phase A of the study will be open to NHS sites around England to take part.

ELIGIBILITY:
Inclusion Criteria:

* Women who are more than 28 weeks pregnant OR up to 9 months post-birth

Exclusion Criteria:

* Outside the limits of the number of weeks pregnant/post birth
* Living outside England
* Refusal to participate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women in the final 3 months of pregnancy or the first 9 months post-birth
Sampling Method: Non-Probability Sample
Enrollment: 2558 (Actual)
Dates: Start 2015-10-19 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
Depression | Retrospective measure since the date of completion of the previous questionnaire
  Measured using the Edinburgh Postnatal Depression Scale

SECONDARY OUTCOMES:
Mental wellbeing | Retrospective measure since the date of completion of the previous questionnaire
  Measured using the short Warwick-Edinburgh Mental Wellbeing Scale
Social functioning | Retrospective measure since the date of completion of the previous questionnaire
  Measured using the Social Provisions Scale
Self-esteem | Retrospective measure since the date of completion of the previous questionnaire
  Measured using the Rosenberg Self-esteem Scale
Further questions assessing health and wellbeing including perceived health, health service utilisation, mother-infant bond and creative participation | Retrospective measure since the date of completion of the previous questionnaire
  A range of self-report questions

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Williamon, PhD, Study Chair — Royal College of Music / Imperial College London
Locations (1):
- Centre for Performance Science, Royal College of Music, London, United Kingdom